CLINICAL TRIAL: NCT04035369
Title: Endophthalmitis Post Intravitreal Injections Comparison EPIIC Trial: Pars Plana Vitrectomy Versus Tap and Inject
Brief Title: Endophthalmitis Post Intravitreal Injections
Acronym: EPIIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPIIC
Record Dates: First submitted 2019-06-19; First posted 2019-07-29 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Endophthalmitis
MeSH Terms: conditions — Endophthalmitis | interventions — Paracentesis

STUDY DESIGN:
Masking Description: Study personnel involved in visual acuity assessments and imaging will be masked to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endophthalmitis Post Intravitreal Injections - TAI (Active Comparator): Patients 18 years and older with presumed infectious endophthalmitis after non-steroid intravitreal injections randomized to TAI
  Interventions: Procedure: Tap and Inject (TAI)
- Endophthalmitis Post Intravitreal Injections - PPV (Active Comparator): Patients 18 years and older with presumed infectious endophthalmitis after non-steroid intravitreal injections randomized to PPV
  Interventions: Procedure: Pars Plana Vitrectomy (PPV)

INTERVENTIONS:
Procedure: Tap and Inject (TAI) — Patients randomized to the TAI group will have a 0.2 mL vitreous specimen collected and a 0.1 mL anterior chamber paracentesis performed to be sent for standard cultures, Gram stain, and sensitivities.
  Intravitreal injection of the following antibiotics: Vancomycin 1.0 mg/0.1 mL, ceftazidime 2.25 mg/0.1 mL (amikacin 400 mcg/0.1 mL instead of Ceftazidime if severe penicillin allergy) and an intravitreal injection of dexamethasone 400 mcg/0.1 mL
  Other Names: TAI
  Arms: Endophthalmitis Post Intravitreal Injections - TAI
Procedure: Pars Plana Vitrectomy (PPV) — Patients randomized to the PPV group will undergo a three-port PPV. The patient should be added to the OR list as an A-case (maximum 6 hours wait) and no intravitreal injection should be performed prior to the surgery. A 0.1 mL aqueous humor simple immediately before the surgery. A 0.2 mL vitreous specimen will be obtained after the sclerotomies are placed. The PPV procedure should be limited to core vitrectomy, air fluid exchange and intravitreal injections (antibiotics and dexamethasone - Vancomycin 1.0 mg/0.1 mL, ceftazidime 2.25 mg/0.1 mL or amikacin 400 mcg/0.1 mL instead of Ceftazidime if severe penicillin allergy and an intravitreal injection of dexamethasone 400 mcg/0.1 mL). Other tamponades such as silicone oil should be avoided if possible. The PPV will then be completed by the surgeon and the vitreous specimen will be sent for standard cultures, Gram stain, and sensitivities.
  Other Names: PPV
  Arms: Endophthalmitis Post Intravitreal Injections - PPV

SUMMARY:
Intravitreal injection (IVI) is an ophthalmological procedure used worldwide to treat ocular conditions. Its use has been steadily increasing for several years, because this method of drug delivery minimizes systemic exposure and allows for intraocular drug levels not achievable through systemic or topical drug administration. IVI of agents such as anti-vascular endothelial growth factor (anti-VEGF) or corticosteroids are efficacious for several retinal diseases, including age-related macular degeneration, macular edema due to retinal vein occlusion or diabetic macular edema, and uveitis, among others. But IVIs are not without their risk of complications and the most feared of which is infectious endophthalmitis, which can occur following intravitreal injections and has potentially devastating visual consequences, including loss of vision and/or the eye itself. Although endophthalmitis´s incidence ranges from 0-0.2% per infection, the cumulative risk for patients under sequential treatment may equate to more than 1% after 2 years of treatment. Endophthalmitis management following IVIs generally consists of a vitreous tap and inject (TAI) and/or a pars plana vitrectomy (PPV) with intravitreal injection of antibiotics. However, there is no consensus on the optimal treatment of IVI-related endophthalmitis. Thus, an established treatment protocol for IVI-related endophthalmitis is warranted to optimize patient outcomes.

The aim of this study is to determine whether PPV or TAI is superior for the treatment of IVI-related endophthalmitis.

DETAILED DESCRIPTION:
Background The use of intravitreal injections (IVIs) has been steadily increasing for several years, because this method of drug delivery minimizes systemic exposure and allows for intraocular drug levels not achievable through systemic or topical drug administration. Intravitreal injection (IVI) of agents such as anti-vascular endothelial growth factor (anti-VEGF) or corticosteroids are efficacious for several retinal diseases, including age-related macular degeneration, macular edema due to retinal vein occlusion or diabetic macular edema, and uveitis, among others. But IVIs are not without their risk of complications and the most feared of which is infectious endophthalmitis. Although endophthalmitis´s incidence ranges from 0-0.2% per infection, the cumulative risk for patients under sequential treatment may equate to more than 1% after 2 years of treatment. Endophthalmitis management following IVIs generally consists of a vitreous tap and inject (TAI) and/or a pars plana vitrectomy (PPV) with intravitreal injection of antibiotics. However, there is no consensus on the optimal treatment of IVI-related endophthalmitis. Thus, an established treatment protocol for IVI-related endophthalmitis is warranted to optimize patient outcomes.

Objectives and Innovation The aim of this study is to determine whether PPV or TAI is superior for the treatment of IVI-related endophthalmitis. The primary objective is to compare final visual acuity (VA) between treatment regimens at 12-months post-treatment. Secondary objectives include subgroup analysis between patients of varying VAs and demographic variables, aqueous humor analysis, comparison of complications and/or need for retreatment, and comparison of anatomic outcomes by autofluorescence, optical coherence tomography (OCT), and OCT angiography (OCTA) imaging.

Methods Consenting patients 18 years and older with presumed infectious endophthalmitis after non-steroid intravitreal injections will undergo stratified block randomized into the PPV or TAI intervention group based on their baseline VA in the study eye. Patient demographics will be collected and a standard ocular examination at baseline will be performed.

Randomization Stratified block randomization (block size = 4) will be used to randomize patients into one of the two interventions according to baseline visual acuity in the study eye (worse than or equal to hand motions and counting fingers or worse) A computer-generated block randomization design will be used to create the randomization list, which will be uploaded to the randomization system (RedCap). Once a patient has consented and been enrolled in the study, the local study coordinator will access the randomization system to enter the patient's assigned study ID and visual acuity status. The treatment group assignment will then be displayed by randomization system to the study coordinator who will inform the recruiting physician.

Masking Study personnel involved in visual acuity assessments and imaging will be masked to group assignment.

Screening Procedures

Patients will be screened by the investigator in the same manner as standard patients. The tests to be performed are typically used for diagnosis and follow-up of endophthalmitis. At each visit (unless indicated otherwise), patients will undergo:

* Best-corrected Snellen visual acuity assessment
* Slip-lamp examination
* Tonometry
* Fundoscopy
* B-scan ultrasound (US) at baseline if the fundus cannot be visualized

Assessment and Procedures

In addition to the above screening procedures, a baseline patient evaluation will be performed that will include thorough documentation of the patient's medical and ocular history. The following will also be performed for each enrolled participant (note that study procedures that are in addition to standard of care have been marked with an asterisk*):

* *ETDRS visual acuity measured at baseline, 3 months, 6 months, and 12 months: the Early Treatment of Diabetic Retinopathy Study (ETDRS) defined a method of visual acuity assessment that has become the gold standard for use in eye research studies. No additional risk is associated with performing ETDRS VA measurements.

  * If no letters can be read at 4 m with an ETDRS chart, the ability to count fingers will be tested at 1 m
  * If unable to count fingers, vision will be tested for the ability to recognize hand motions in which the opposite eye will be occluded and a light source will be directed from behind the patient to the examiner's hand that will be stationary or moved at one motion per second in a horizontal or vertical direction at a distance of 60 cm from the eye. The patient will then identify the direction of the examiner's hand. This procedure will be repeated five times and hand-motion VA will be considered present if the patient is able to identify the examiner's action on at least four of the presentations.
  * Light perception (LP) will be tested at 0.9 m with an indirect ophthalmoscope at maximum intensity
* *Visual Function Questionnaire 25 (VFQ-25) administered at baseline, 3 months, 6 months, and 12 months: a questionnaire developed by the National Eye Institute29-31 to measure visual function in 11 domains encompasses areas of general vision, ocular pain, near activities, distance activities, vision-specific social functioning, vision-specific mental health, vision-specific role difficulties, vision-specific dependency, driving, color vision, and peripheral vision. No additional risk is associated with administering the VFQ-25 Questionnaire.
* *The 36-Item Short-Form Survey (SF-36) administered at baseline, 1 month and 1 year: It is a patient-reported survey of patient health. No additional risk is associated with administering the 36-Item Short-Form Questionnaire.
* Fundus autofluorescence at 3 months (mandatory)
* Optos photographs at 3 months and 12 months (mandatory)
* OCT 5 HD-line images at 3 months, 6 months and 12 months (mandatory)
* OCT-A images at 3 months and 12 months (optional)
* Anterior chamber paracentesis to obtain a 0.1 mL aqueous humour sample prior to treatment: this sample will be sent for standard cultures, Gram stain, and sensitivities.
* Vitreous samples to obtain a 0.2mL vitreous sample prior to treatment: this sample will be sent for standard cultures, Gram stain, and sensitivities.
* Cataract surgery: may be considered for patients who subsequently develop visually significant cataracts as a result of the intervention (likely needed for those in the PPV group)

  * this will be assessed at 6 months and cataract surgery will be offered if the cataract is visually significant
  * if the patient declines, cataracts will be re-assessed at 9 months and cataract surgery will be re-offered

Pars Plana Vitrectomy Group Patients randomized to the PPV group will undergo a three-port PPV. The patient should be added to the OR list as an A-case (maximum 6 hours wait) and no intravitreal injection should be performed prior to the surgery. A 0.1 mL aqueous humor simple immediately before the surgery. A 0.2 mL vitreous specimen will be obtained after the sclerotomies are placed. The PPV procedure should be limited to core vitrectomy, air fluid exchange and intravitreal injections (antibiotics and dexamethasone). Other tamponades such as silicone oil should be avoided if possible. The PPV will then be completed by the surgeon and the vitreous specimen will be sent for standard cultures, Gram stain, and sensitivities.

Tap and Inject Group Patients randomized to the TAI group will have a 0.2 mL vitreous specimen collected and a 0.1 mL anterior chamber paracentesis performed to be sent for standard cultures, Gram stain, and sensitivities.

Medications

Following the PPV or tap, each patient will receive the following empirical therapy:

* Intravitreal injection of antibiotics

  * Vancomycin 1.0 mg/0.1 mL
  * Ceftazidime 2.25 mg/0.1 mL
  * Amikacin 400 mcg/0.1 mL instead of Ceftazidime if severe penicillin allergy
* Intravitreal injection of dexamethasone 400 mcg/0.1 mL
* Oral moxifloxacin 400 mg OD for 10 days. (start as soon as possible)
* Topical moxifloxacin q1h x 48 hours post-treatment, then tapered according to treating physician's standard regimen
* Topical Prednisolone 1%: q1h x 48 hours post-treatment, then tapered according to treating physician's standard regimen
* Any mydriatic agent typically used by the treating physician and according to their standard regimen

Rescue Treatment and Risk Management For patients in the TAI group, PPV and reinjection of intravitreal antibiotics can be considered if the infection worsens after the initial intervention. Patients in the PPV group can be considered for repeat PPV and reinjection of intravitreal antibiotics if the infection worsens after the initial intervention as well. The final decision for retreatment will be at the physician's discretion and what they judge to be in the patient's best interest.

Safety Monitoring Plan A Data and Safety Monitoring Board (DSMB) will meet annually. Voting members of the DSMB will be independent of the trial. A written report containing the current status of the trial, performance and data quality, interim outcome data will be sent to DSMB members by the Coordinating Center to allow sufficient time for the DSMB members to review the report prior to the meeting. This report will address any specific concerns about the conduct of the trial.

Also, the local principal investigator (LPI) at each site will meet weekly with study team members to review the progress of the study. Furthermore, to ensure all members are performing their roles in accordance with required Research Ethics Board requirements, the LPI will randomly check on the study coordinators and participants.

The TAI and PPV interventions will be performed or supervised by qualified ophthalmologists. Patients will be made fully aware of the risk and benefits of the procedures. Patients will be assessed pre- and post-intervention for any adverse events, and will be closely monitored throughout the study. Complications will be managed by the staff ophthalmologist and other necessary eye clinic staff.

Statistical Analysis

Data will be upload on electronic case report form, provided by the Applied Health Research Centre ("AHRC") of St. Michael's Hospital.

Continuous variables will be reported as means with standard deviations or median with minimum and maximum values, and will be compared using T-tests or Mann-Whitney U tests. Categorical measures will be reported as counts and percentages, and will be compared using Chi-squared tests or Fisher's Exact test.

ETDRS visual acuity and VFQ-25 scores at 3 months, 6 months, and 12 months, will be compared between groups using an independent t-test. Linear regression models will be used to determine the relationship between various patient-related baseline factors and final ETRDS VA at 12 months within each group.

Coefficients with 95% confidence intervals will be reported. A p-value of 0.05 will be considered for statistical significance. Data will be analyzed using SPSS (SPSS Inc., Chicago, IL).

Sample Size A sample size calculation was performed in relation to the primary outcome to detect a difference in ETDRS VA of 10 letters (2-line difference) between groups. With a study powered to 90%, an alpha of 0.05, and standard deviation of 25 letters, this results in a sample size of 278 patients. Assuming a 10% drop out rate, 310 patients are required in total (155 patients in each group).

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years and older
* Intravitreal injections other than intravitreal steroids within the last 2 weeks
* Diagnosed with presumed infectious endophthalmitis: patients presenting with vision loss and hypopyon
* Visual acuity of light perception or better
* Safety concern by the treating physician for patients enrolled in the study. That is to say, if the physician feels a patient's outcomes would be better with one intervention over the other, this patient should not be enrolled in the study.

Exclusion Criteria:

* Prior intraocular surgery in the study eye within the last 3 months
* Prior penetrating ocular trauma
* Bleb or prior glaucoma filtration surgery in the study eye
* Patients with other ocular conditions limiting vision in the study eye other than the retinal pathology for which they receive intravitreal injections for e.g. anterior segment pathology, retinal detachments, end-stage glaucoma
* Previous vitreo-retinal surgery.
* Unwilling or unable to follow or comply with all study-related procedures or sign consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Visual acuity outcomes | 12 months
  To compare visual acuity (VA) measured by Early Treatment of Diabetic Retinopathy Study (ETDRS) testing between PPV and TAI for treatment of endophthalmitis at 12-months post-treatment
  We hypothesize that PPV will be superior to TAP in terms of ETDRS visual outcomes at the 12-month time point.

SECONDARY OUTCOMES:
Early visual acuity outcomes | 3 and 6 months
  Compare ETDRS VA between treatment modalities at 3 and 6 months.
Visual outcomes related to baseline visual acuity | 3, 6 and 12 months
  Subgroup analysis between treatment groups for patients with different pre-endophthalmitis baseline vision based on vision thresholds of 20/40 or better, 20/50 to 20/200, and 20/400 to CF, performed at 3 months, 6 months, and 12 months: the most recently recorded pre-endophthalmitis Snellen visual acuity will be obtained from patient charts and used as the pre-endophthalmitis vision baseline
The Visual Function Questionnaire (VFQ-25) outcomes | 3, 6 and 12 months
  Compare scores from the Visual Function Questionnaire (VFQ-25) between treatment modalities at 3 months, 6 months, and 12 months. The VFQ-25 consists of a base set of 25 vision targeted questionnaire. All items are scored so that a high score represents better functioning. Each item is then converted to a 0 to 100 scale so that the lowest and highest possible scores are set at 0 and 100 points, respectively. In this format scores represent the achieved percentage of the total possible score, e.g. a score of 50 represents 50% of the highest possible score.
The 36-Item Short-From Survey (SF-36) | Baseline, 1 month and 12 months
  Compare scores from the 36-Item Short-From Survey (SF-36) between treatment modalities at baseline, 1 month and 1 year. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
Number of participants with treatment-related adverse events as assessed by OCT | 3, 6 and 12 months
  The participants will be evaluated as "Yes" or "No" to de following OCT findings: 1- Cystoid macular edema (CME); 2- Subretinal fluid (SRF); 3- Intraretinal fluid (IRF); 4-Epiretinal membrane (ERM); 5-Macular hole (MH)
Number of participants with treatment-related adverse events as assessed by Optos retinal photos | 3 and 12 months
  The participants will be evaluated as "Yes" or "No" to de following Optos Photos: 1-Retina status attached; 2-Epiretinal membrane (ERM); 3-Cystoid macular edema (CME); 4-Retinal Ischemia; 5-Retinal hemorrhages
Number of participants with treatment-related adverse events as assessed by Autofluorescence (AF) images | 3 months
  The participants will be evaluated as "Yes" or "No" to de following Autofluorescence: 1-Retina status attached; 2-Retinal lesion activity; 3-Retinal scar
Complications and retreatment | 12 months
  Comparison of complications and/or need for retreatment following each intervention
Aqueous humor and vitreous sample Culture | Baseline
  Standard cultures: 1=Coagulase-negative staphylococci; 2=Staphylococcus Aureus; 3= Staphylococcus Epidermidis; 4=Streptococcus Pneumoniae; 5=H. influenzae; 6=Other; 7=No growth
Aqueous humor and vitreous sample Gram stain | Baseline
  Gram stain: ( ) positive; ( ) negative; ( ) fungi; ( ) organisms not detected
Aqueous humor and vitreous sample Sensitivities | Baseline
  Antibiotics sensitivities: ( ) vancomycin; ( )ceftazidime; ( ) gatifloxacine; ( ) ofloxacin ( ) polymyxin; ( ) bacitracin; ( ) trimethoprim; ( ) cefazolin; ( ) ceftriaxone;
Changes in visual acuity | 3, 6 and 12 months
  Analysis of the changes in the visual acuity during the study
Recovery to the pre-endophthalmitis visual acuity | 3, 6 and 12 months
  Analysis in patients recovering the pre-endophthalmitis visual acuity and timing (in months) from treatment to recovery.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Michael's Hospital Eye Clinic, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chaudhary KM, Romero JM, Ezon I, Fastenberg DM, Deramo VA. Pars plana vitrectomy in the management of patients diagnosed with endophthalmitis following intravitreal anti-vascular endothelial growth factor injection. Retina. 2013 Jul-Aug;33(7):1407-16. doi: 10.1097/IAE.0b013e3182807659. PMID 23492945
- [Background] Xu K, Chin EK, Bennett SR, Williams DF, Ryan EH, Dev S, Mittra RA, Quiram PA, Davies JB, Parke DW 3rd, Johnson JB, Cantrill HL, Almeida DRP. Endophthalmitis after Intravitreal Injection of Vascular Endothelial Growth Factor Inhibitors: Management and Visual Outcomes. Ophthalmology. 2018 Aug;125(8):1279-1286. doi: 10.1016/j.ophtha.2018.01.022. Epub 2018 Feb 21. PMID 29477689
- [Background] Results of the Endophthalmitis Vitrectomy Study. A randomized trial of immediate vitrectomy and of intravenous antibiotics for the treatment of postoperative bacterial endophthalmitis. Endophthalmitis Vitrectomy Study Group. Arch Ophthalmol. 1995 Dec;113(12):1479-96. PMID 7487614
- [Background] Haddock LJ, Ramsey DJ, Young LH. Complications of subspecialty ophthalmic care: endophthalmitis after intravitreal injections of anti-vascular endothelial growth factor medications. Semin Ophthalmol. 2014 Sep-Nov;29(5-6):257-62. doi: 10.3109/08820538.2014.959616. PMID 25325851
- [Background] Moss JM, Sanislo SR, Ta CN. Antibiotic susceptibility patterns of ocular bacterial flora in patients undergoing intravitreal injections. Ophthalmology. 2010 Nov;117(11):2141-5. doi: 10.1016/j.ophtha.2010.02.030. Epub 2010 Jun 18. PMID 20561687
- [Result] Irigoyen C, Ziahosseini K, Morphis G, Stappler T, Heimann H. Endophthalmitis following intravitreal injections. Graefes Arch Clin Exp Ophthalmol. 2012 Apr;250(4):499-505. doi: 10.1007/s00417-011-1851-1. Epub 2011 Nov 3. PMID 22048244